CLINICAL TRIAL: NCT06426407
Title: Vasopressin Hemodynamic Response as a Septic Shock Subphenotype Indicator
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Seth Bauer, Principal Investigator, The Cleveland Clinic
Other Study IDs: 21-047
Record Dates: First submitted 2024-02-16; First posted 2024-05-23 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Shock, Septic
MeSH Terms: conditions — Shock, Septic | interventions — Vasopressins; Arginine Vasopressin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood collected into EDTA test tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vasopressin plus norepinephrine: Patients with septic shock ordered vasopressin as an adjunct to norepinephrine
  Interventions: Drug: Vasopressin
- Norepinephrine: Active control cohort of patients with septic shock who are only receiving norepinephrine

INTERVENTIONS:
Drug: Vasopressin — Fixed dosage vasopressin ordered as an adjunctive vasopressor to norepinephrine
  Other Names: antidiuretic hormone (ADH); arginine vasopressin (AVP)
  Groups: Vasopressin plus norepinephrine

SUMMARY:
The goal of this observational study is to learn about blood pressure response to the vasopressor drug vasopressin in people with septic shock.

The main questions it aims to answer are:

* Are the levels of molecules showing communication between cells different between people whose blood pressure improves and people whose blood pressure does not improve when given a vasopressor medication?
* Are measurements found on echocardiography (heart ultrasound) different between people whose blood pressure improves and people whose blood pressure does not improve when given a vasopressor medication?
* Are measurements of blood oxygen in tissues just below the skin different between people whose blood pressure improves and people whose blood pressure does not improve when given a vasopressor medication?

Participants will be asked to contribute one or two blood samples. Participants who are ordered the drug vasopressin will contribute two blood samples. Both samples will be about two tablespoons for a total of about four tablespoons. One sample will be drawn before starting vasopressin infusion and the second sample will be drawn between one and six hours after starting the vasopressor drug infusion. At the same time points, advanced echocardiography pictures and measurements of oxygen in tissues from a sensor placed on one of the hands will be taken. Participants who are not ordered the drug vasopressin and only ordered the drug norepinephrine will contribute only one blood sample. At the time the sample is collected, advanced echocardiography pictures and measurements of oxygen in tissues from a sensor placed on one of the hands will be taken. This research also involves analyzing data obtained during the participant's hospital stay.

DETAILED DESCRIPTION:
Septic shock mortality remains high at 33% in North America; current clinical predictors of poor outcomes in septic shock are suboptimal. In addition to antibiotics and intravenous fluids, vasoactive agents are initiated to restore effective tissue perfusion. Norepinephrine (NE) is the recommended first-line vasopressor, but adjunctive arginine vasopressin is used in over one-third of patients to improve blood pressure or decrease NE dosage. However, less than half of vasopressin recipients have a clinically-apparent hemodynamic response (defined as a decrease in NE dosage at 6 hours after vasopressin initiation). Vasopressors, particularly norepinephrine, are known to be immune modulators. Further, each vasopressor has its own unique effect on a patient's hemodynamic profile as assessed by echocardiography and microcirculation measurements. In the current study, the investigators seek to clarify the link between vasopressin, immune response, hemodynamic profile, and microcirculatory measurments. The central goal of this proposal is to identify "vasopressin response" as an easily-identifiable bedside indicator of a distinct septic shock subphenotype.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old)
* Septic shock (as defined by Sepsis-3)
* Receiving norepinephrine
* Admitted to a medical, surgical, NeuroSciences, or mixed intensive care unit
* Central venous catheter in place
* Ordered fixed-dose vasopressin as an adjunct to norepinephrine by the primary care team (unless in active control cohort)

Exclusion Criteria:

* Vasopressin ordered for an indication other than septic shock
* Vasopressin initiated at another institution
* Receiving a primary vasopressor other than norepinephrine (eg, phenylephrine)
* Positive test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) within the preceding 28 days
* Blood hemoglobin concentration <7 g/dL
* Primary treatment team determines that vasopressin initiation is emergent
* Patient or their legal authorized representative opts to not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with septic shock are eligible for this study. Patients ordered vasopressin as an adjunct to norepinephrine as part of routine care comprise the primary cohort of interest. An active control cohort of patients who are only receiving norepinephrine will also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Ratio of plasma interleukin-10 (IL-10) to tumor necrosis factor-α (TNF-α) | Baseline (before vasopressin initiation and within 45 minutes of order placement).
  Compare baseline ratio of plasma concentrations of interleukin-10 (IL-10) to tumor necrosis factor-α (TNF-α) in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | Baseline (before vasopressin initiation and within 45 minutes of order placement).
  Compare baseline left ventricular ejection fraction (LVEF) in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Ratio of ratio of arterial elastance (Ea) to left ventricular end-systolic elastance (Ees) | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare left ventricular-arterial coupling (ratio of arterial elastance [Ea] to left ventricular end-systolic elastance [Ees]) over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Lipopolysaccharide-stimulated monocyte TNF-α secretion | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare lipopolysaccharide-stimulated monocyte TNF-α secretion over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Monocyte adhesion | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare monocyte adhesion over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Plasma renin concentration | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare plasma renin concentration over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Plasma angiopoietin-2 concentration | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare plasma angiopoietin-2 concentration over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
StO2 recovery slope (%/min) | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare tissue oxygenation (StO2) recovery slope, during the reperfusion phase of a vascular occlusion test (VOT), over time between vasopressin responders vs non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Difference in StO2 (%) | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare the difference between maximum tissue oxygenation (StO2) and minimum StO2, during the reperfusion phase of a vascular occlusion test (VOT), over time between vasopressin responders vs non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.

OTHER OUTCOMES:
Plasma interleukin-1β (IL-1β) concentration | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare plasma interleukin-1β (IL-1β) concentration over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Plasma interleukin-6 (IL-6) concentration | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare plasma interleukin-6 (IL-6) concentration over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Plasma interferon-gamma (IFN-γ) concentration | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare plasma interferon-gamma (IFN-γ) concentration over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Plasma C-X-C motif chemokine ligand 10 (CXCL10, also known as interferon gamma-induced protein 10 [IP-10]) concentration | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare plasma C-X-C motif chemokine ligand 10 (CXCL10, also known as interferon gamma-induced protein 10 [IP-10]) concentration over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Plasma granulocyte-colony stimulating factor (G-CSF) concentration | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare plasma granulocyte-colony stimulating factor (G-CSF) concentration over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Plasma E-selectin concentration | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare plasma E-selectin concentration over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Plasma vasopressin concentration | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Evaluate the association of plasma vasopressin concentration with ratio of plasma interleukin-10 (IL-10) to tumor necrosis factor-α (TNF-α) over time. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Plasma copeptin concentration | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare plasma copeptin concentration over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Left ventricular ejection fraction (LVEF) change | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare left ventricular ejection fraction (LVEF) over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Stroke volume (SV) by echocardiography | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare stroke volume (SV) over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Tricuspid annular plane systolic excursion (TAPSE) | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare tricuspid annular plane systolic excursion (TAPSE) over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Tricuspid annular systolic plane velocity (TAPSV, also known as RV S') | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare tricuspid annular systolic plane velocity (TAPSV, also known as RV S') over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Venous-arterial carbon dioxide tension gradient (Pva-CO2) | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare venous-arterial carbon dioxide tension gradient (Pva-CO2) over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Central venous oxygen saturation (ScvO2) | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare central venous oxygen saturation (ScvO2) over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Dynamic arterial elastance (Eadyn, the ratio of pulse pressure variation to stroke volume variation) | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare dynamic arterial elastance (Eadyn) over time in vasopressin responders vs. non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Baseline tissue oxygenation (StO2) | Baseline (before vasopressin initiation and within 45 minutes of order placement).
  Compare baseline tissue oxygenation (StO2) over time between vasopressin responders vs non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Tissue oxygenation (StO2) deperfusion slope | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare tissue oxygenation (StO2) deperfusion slope, during a vascular occlusion test, over time between vasopressin responders vs non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Minimum tissue oxygenation (StO2) | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare minimum tissue oxygenation (StO2), during a vascular occlusion test, over time between vasopressin responders vs non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Tissue oxygenation (StO2) area under the curve (AUC) | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare tissue oxygenation (StO2) area under the curve (AUC), during a vascular occlusion test, over time between vasopressin responders vs non-responders. The active control cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Capillary refill time (CRT) | Baseline (before vasopressin initiation and within 45 minutes of order placement) through one to six hours after vasopressin initiation.
  Compare capillary refill time (CRT) over time between vasopressin responders vs non-responders. The active control of cohort of patients who are only receiving norepinephrine will serve as a control for this analysis.
Clinical trajectory | Baseline (before vasopressin initiation and within 45 minutes of order placement) through the sooner of intensive care unit discharge or 14 days.
  Compare the ordinal outcome clinical trajectory (comprised of rapid recovery, chronic critical illness, and early recovery) between vasopressin responders vs. non-responders.
Intensive care unit length of stay | Baseline (before vasopressin initiation and within 45 minutes of order placement) through intensive care unit discharge.
  Compare intensive care unit length of stay in vasopressin responders vs. non-responders.
Incidence of in-hospital mortality | Baseline (before vasopressin initiation and within 45 minutes of order placement) through hospital discharge.
  Compare the incidence of hospital mortality in vasopressin responders vs. non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Bauer, PharmD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be available through reasonable request to the study principal investigator and completion of a data use agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study data will become available at the time of initial manuscript publication and remain available for 5 years after initial manuscript publication.
Access Criteria: Individual participant data may be available through reasonable request to the study principal investigator and completion of a data use agreement.